CLINICAL TRIAL: NCT05980949
Title: Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of KarXT in Subjects With Psychosis Associated With Alzheimer's Disease (ADEPT-3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0028; CN012-0028 (Other: Bristol-Myers Squibb Protocol ID); KAR-033 (Other: Karuna Pharmaceuticals Protocol ID); 2023-504151-27 (Other: EU CTR)
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Psychosis Associated With Alzheimer's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental): Xanomeline and Trospium Chloride Capsules
  Interventions: Drug: KarXT

INTERVENTIONS:
Drug: KarXT — KarXT 20/2 mg TID (total daily dose [TDD] 60/6 mg) KarXT 30/3 mg TID (TDD 90/9 mg) KarXT 40/4 mg TID (TDD 120/12 mg) KarXT 50/5 mg TID (TDD 150/15 mg) KarXT 66.7/6.67 mg TID (TDD 200/20 mg)

SUMMARY:
This is a Phase 3 global, multicenter, 52-week, open-label extension (OLE) rollover study for subjects completing study CN012-0026, CN012-0027 or CN012-0056. Subjects (randomized or non-randomized) who complete the 38-week CN012-0026 study, 14-week CN012-0027 study or 14-week CN012-0056 study will be eligible to enroll in CN012-0028. The primary objective of the study is to assess the long-term safety and tolerability of KarXT in subjects with psychosis associated with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed study CN012-0026, CN012-0027 or CN012-0056.
* Subject was aged 55 to 90 years, inclusive, at the time of enrollment into the parent CN012-0026, CN012-0027 or CN012-0056 study.
* Can understand the nature of the study and protocol requirements and provide a signed informed consent or, if deemed not competent to provide informed consent, the subject's legally acceptable representative must provide informed consent, and the subject must provide informed assent before any study assessments are performed.
* At entry into this study, or any time during the study, if a subject needs to relocate from home or residential assisted-living facility to a nursing home facility, the Sponsor/Medical Monitor must approve the subject's participation in the study.
* Have an identified or proxy caregiver (spends approximately 10 hours/week with the subject).

Exclusion Criteria:

* Significant or severe medical conditions that, in the opinion of the Investigator, could jeopardize the safety of the subject, ability to complete or comply with the study procedures or validity of the study results.
* Clinically significant abnormalities, including any finding(s) from the ECG, laboratory tests, physical examination, or vital signs, at the EOT visit of Study CN012-0026, CN012-0027 or CN012-0056 that the Investigator, in consultation with the Medical Monitor, are considered to jeopardize the safety of the subject.
* Subjects participating in another investigational drug or device study or planning on participating in another clinical study during the duration of CN012-0028.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-09-07 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From initial dose through 14 days after the final dose (up to 54 weeks)
  The number and percentage of participants with TEAEs will be determined

SECONDARY OUTCOMES:
Incidence of serious TEAEs | From initial dose through 14 days after the final dose (up to 54 weeks)
  The number and percentage of participants with serious TEAEs will be determined
Incidence of TEAEs leading to withdrawal | From initial dose through 14 days after the final dose (up to 54 weeks)
  The number and percentage of participants with TEAEs leading to withdrawal will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (411):
- United States (142):
  - Local Institution - 1029, Homewood, Alabama
  - Local Institution - 1-13H98LK9, Chandler, Arizona
  - Local Institution - 1227, Chandler, Arizona
  - Local Institution - 1116, Chandler, Arizona
  - Local Institution - 1217, Phoenix, Arizona
  - Local Institution - 1044, Phoenix, Arizona
  - Local Institution - 1220, Scottsdale, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Local Institution - 1-141NO1DG, Chino, California
  - Local Institution - 1001, Costa Mesa, California
  - Local Institution - 1151, Encino, California
  - Local Institution - 1033, Encino, California
  - Local Institution - 1031, Irvine, California
  - Local Institution - 1230, Lakewood, California
  - Local Institution - 1142, Lancaster, California
  - Local Institution - 1117, Los Alamitos, California
  - USC - The Memory and Aging Center (MAC) - Alzheimer Disease Research Center (ADRC), Los Angeles, California
  - Local Institution - 1228, Orange, California
  - SC3 Research - Pasadena - 960 E. Green St, Pasadena, California
  - Local Institution - 1213, Rancho Cucamonga, California
  - California Neuroscience Research - CenExel - PPDS, Sherman Oaks, California
  - Local Institution - 1007, Walnut Creek, California
  - Local Institution - 1014, Colorado Springs, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Local Institution - 1013, Stamford, Connecticut
  - Local Institution - 1225, Atlantis, Florida
  - Local Institution - 1011, Boca Raton, Florida
  - Local Institution - 1020, Bonita Springs, Florida
  - Local Institution - 1015, Bradenton, Florida
  - Local Institution - 1156, Clermont, Florida
  - K2 Medical Research - Winter Garden, Clermont, Florida
  - JY Research Institute Inc, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Local Institution - 1224, Deerfield Beach, Florida
  - Local Institution - 1162, Delray Beach, Florida
  - Integrity Clinical Research, LLC - 8000 NW 21st St, Doral, Florida
  - Betancourt Research Services, Doral, Florida
  - Local Institution - 1165, Fort Myers, Florida
  - Superior Associates in Research LLC, Hialeah, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - New Life Medical Research Center -3750 W 16th Ave, Hialeah, Florida
  - Local Institution - 1046, Hialeah, Florida
  - Las Mercedes Medical Research - 4440 West 16th Ave, Hialeah, Florida
  - Local Institution - 1-13JED81K, Hialeah, Florida
  - Local Institution - 1237, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Nexus Clinical Research Center- NRC, Homestead, Florida
  - Local Institution - 1145, Homestead, Florida
  - Coral Clinic Research, Homestead, Florida
  - Homestead Associates in Research Inc-30328 Old Dixie Hwy, Homestead, Florida
  - Local Institution - 1127, Largo, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - Local Institution - 1146, Maitland, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Angels Clinical Research Institute - Miami, Miami, Florida
  - Local Institution - 1005, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Wellness Research Center Inc - Miami, Miami, Florida
  - A & D Doctor Center, Miami, Florida
  - Floridian Neuroscience Institute-1901 SW 1 St, Miami, Florida
  - Local Institution - 1010, Miami, Florida
  - MedOne Clinical Research LLC, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - My Community Research Center, Inc - 7480 Bird Rd, Miami, Florida
  - Future Care Solution LLC, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Local Institution - 1053, Miami, Florida
  - Local Institution - 1006, Miami, Florida
  - Dade Research Center - Miami FL - 7600 SW 87th Ave, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - US Associates in Research Inc, Miami, Florida
  - Serenity Research Center, Miami, Florida
  - IMIC LLC- 9380 SW 150th Str, Miami, Florida
  - New Gen Health, Miami, Florida
  - Floridian Research Institute-1021 Ives Dairy Rd, Miami, Florida
  - High Quality Research, Miami, Florida
  - Coral Research Clinic & Coral Diagnostic Center, Miami, Florida
  - ONHEALTH Research Center, Miami, Florida
  - New Med Research, Miami Gardens, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - Meridian International Research, Miami Lakes, Florida
  - Local Institution - 1209, Miami Lakes, Florida
  - Ocean Blue Medical Research Center Inc, Miami Springs, Florida
  - Local Institution - 1246, Naples, Florida
  - Local Institution - 1212, Ocoee, Florida
  - Local Institution - 1101, Okeechobee, Florida
  - Local Institution - 1242, Orlando, Florida
  - Local Institution - 1136, Orlando, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Local Institution - 1012, Pensacola, Florida
  - Local Institution - 1137, Port Orange, Florida
  - Local Institution - 1205, Port Orange, Florida
  - Local Institution - 1008, St. Petersburg, Florida
  - Cordova Research Institute- Sweetwater, Sweetwater, Florida
  - Local Institution - 1041, Tampa, Florida
  - Guardian Angel Research - ClinEdge - PPDS, Tampa, Florida
  - Angels Clinical Research Institute Tampa - Palm Springs - PPDS, Tampa, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Local Institution - 1040, The Villages, Florida
  - Local Institution - 1131, Viera, Florida
  - Premiere Research Institute at Palm Beach Neurology, PA, West Palm Beach, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Local Institution - 1161, Decatur, Georgia
  - Local Institution - 1037, Berwyn, Illinois
  - Local Institution - 1148, Elgin, Illinois
  - Local Institution - 1114, Marrero, Louisiana
  - Local Institution - 1223, Belmont, Massachusetts
  - Local Institution - 1245, Boston, Massachusetts
  - Local Institution - 1243, North Dartmouth, Massachusetts
  - Local Institution - 1239, Springfield, Massachusetts
  - Local Institution - 1-146Y4PVY, Bloomfield Township, Michigan
  - Local Institution - 1139, Rochester Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Bio Behavioral Health - 20 Hospital Dr, Toms River, New Jersey
  - Local Institution - 1202, Toms River, New Jersey
  - Local Institution - 1018, Manhasset, New York
  - Local Institution - 1017, New York, New York
  - Local Institution - 1034, Stony Brook, New York
  - Local Institution - 1231, Syracuse, New York
  - Local Institution - 1240, Syracuse, New York
  - Five Towns Neurology PC -Woodmere - 923 Broadway, Woodmere, New York
  - Local Institution - 1221, Greensboro, North Carolina
  - Local Institution - 1214, Matthews, North Carolina
  - Local Institution - 1215, Morehead City, North Carolina
  - Local Institution - 1201, Columbus, Ohio
  - Local Institution - 1122, Dayton, Ohio
  - Local Institution - 1249, Shaker Heights, Ohio
  - Local Institution - 1016, Oklahoma City, Oklahoma
  - Local Institution - 1218, Providence, Rhode Island
  - Local Institution - 1035, Charleston, South Carolina
  - Local Institution - 1211, Nashville, Tennessee
  - Horizon Clinical Research: Gill Neuroscience, Cypress, Texas
  - Local Institution - 1121, DeSoto, Texas
  - Local Institution - 1208, El Paso, Texas
  - Local Institution - 1022, Flower Mound, Texas
  - Local Institution - 1036, Frisco, Texas
  - Clinical Trial Network - 7080 Southwest Fwy, Houston, Texas
  - Local Institution - 1238, Plano, Texas
  - Local Institution - 1210, San Antonio, Texas
  - Local Institution - 1134, Stafford, Texas
  - Local Institution - 1241, Arlington, Virginia
- Argentina (9):
  - Local Institution - 5004, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5009, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5005, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5001, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5008, Rosario, Santa Fe Province
  - Local Institution - 5002, Buenos Aires
  - Local Institution - 5006, Buenos Aires
  - Local Institution - 5003, Córdoba
  - Local Institution - 5007, San Rafael
- Belgium (7):
  - Local Institution - 2806, Jette, Brussels Capital
  - Local Institution - 2801, Hasselt, Limburg
  - Local Institution - 2802, Leuven, Vlaams Brabant
  - Local Institution - 2803, Roeselare, West-Vlaanderen
  - Local Institution - 1-13JED87R, Alken
  - Local Institution - 2804, Alken
  - Local Institution - 2805, Kortrijk
- Brazil (13):
  - Local Institution - 1-13J38ZST, Brasília, Federal District
  - Local Institution - 6201, Brasília, Federal District
  - CPQuali Pesquisa Clínica Sao Paulo, São Paulo, São Paulo
  - Local Institution - 1-13J38ZS5, São Paulo, São Paulo
  - Local Institution - 1-13J38ZTW, São Paulo, São Paulo
  - Local Institution - 6206, São Paulo, São Paulo
  - Local Institution - 6207, São Paulo, São Paulo
  - Local Institution - 1-13J38ZSH, São Paulo, São Paulo
  - Clinilive, São Paulo, São Paulo
  - Local Institution - 1-13J38ZRS, São Paulo, São Paulo
  - Local Institution - 1-13J338E3, Rio de Janeiro
  - Ruschel Medicina, Rio de Janeiro
  - Local Institution - 6205, São Paulo
- Bulgaria (8):
  - Medical Center Sveti Naum EOOD, Sofia, Sofia-Grad
  - Local Institution - 4505, Sofia, Sofia-Grad
  - Local Institution - 4502, Sofia, Sofia-Grad
  - Local Institution - 4506, Sofia, Sofia-Grad
  - Medical Center Medconsult Pleven OOD, Pleven
  - Local Institution - 4508, Plovdiv
  - University Multiprofile Hospital For Active Treatment Kanev AD, Rousse
  - Local Institution - 4509, Sofia
- Canada (5):
  - Local Institution - 1-12IRCCNP, Calgary, Alberta
  - Local Institution - 1603, Hamilton, Ontario
  - Local Institution - 1604, Whitby, Ontario
  - Local Institution - 1-12IYJCH7, Montreal, Quebec
  - Local Institution - 1601, Verdun, Quebec
- Chile (3):
  - Biomedica Research Group, Providencia, Santiago Metropolitan
  - Psicomed Estudios Médicos Cía Ltda, Antofagasta
  - Especialidades Medicas L Y S, Las Condes
- China (28):
  - Local Institution - 7007, Hefei, Anhui
  - Local Institution - 7004, Beijing, Beijing Municipality
  - Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality
  - Local Institution - 7025, Beijing, Beijing Municipality
  - Local Institution - 7015, Chongqing, Chongqing Municipality
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Local Institution - 7009, Guangzhou, Guangdong
  - Shenzhen Kangning Hospital, Shenzhen, Guangdong
  - Local Institution - 7014, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Local Institution - 7024, Nanjing, Jiangsu
  - Local Institution - 7023, Zhenjiang, Jiangsu
  - Local Institution - 7012, Nanchang, Jiangxi
  - Shanghai Mental Health Center - PPDS, Shanghai, Shanghai Municipality
  - Local Institution - 7028, Shanghai, Shanghai Municipality
  - Local Institution - 7011, Shanghai, Shanghai Municipality
  - Local Institution - 7026, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Anding Hospital(Tianjin mental Health Center), Tianjin, Tianjin Municipality
  - Local Institution - 7017, Hangzhou, Zhejiang
  - Local Institution - 7010, Hangzhou, Zhejiang
  - Local Institution - 7021, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine - Qingchun Campus, Hangzhou, Zhejiang
  - Local Institution - 7018, Wenzhou, Zhejiang
  - Local Institution - 7027, Changsha
  - Local Institution - 7022, Kunming
- Croatia (6):
  - Klinicki Bolnicki Centar Zagreb, Zagreb, City of Zagreb
  - Local Institution - 1-140R4546, Zagreb, City of Zagreb
  - Local Institution - 4102, Zagreb, City of Zagreb
  - Local Institution - 4103, Zagreb, City of Zagreb
  - Klinika za psihijatriju Vrapce, Zagreb, City of Zagreb
  - Local Institution - 4104, Zagreb, City of Zagreb
- Czechia (5):
  - CLINTRIAL s.r.o., Prague, Praha, Hlavní Mesto
  - Neuroterapie KH, s.r.o Psychiatricka ambulance, Kutná Hora
  - A-SHINE s.r.o., Pilsen
  - Local Institution - 4004, Prague
  - Local Institution - 4006, Rychnov nad Kněžnou
- France (5):
  - Local Institution - 2510, Nice, Alpes-Maritimes
  - Local Institution - 2511, Tours, Indre-et-Loire
  - Local Institution - 2501, Reims, Marne
  - Centre Hospitalier Universitaire Hopitaux de Rouen-1 Rue de Germont, Rouen, Seine-Maritime
  - Local Institution - 2513, Toulouse
- Germany (8):
  - Local Institution - 2401, Böblingen, Baden-Wurttemberg
  - Local Institution - 2407, Böblingen, Baden-Wurttemberg
  - Local Institution - 2403, Bayreuth, Bavaria
  - Local Institution - 1-13JED8BL, Erbach im Odenwald, Hesse
  - Local Institution - 2402, Homburg, Saarland
  - Local Institution - 2404, Erbach im Odenwald
  - Local Institution - 1-13JED842, Frankfurt am Main
  - Local Institution - 2405, Frankfurt am Main
- Greece (7):
  - Local Institution - 4805, Athens, Attica
  - Local Institution - 4803, Athens, Attica
  - Local Institution - 4802, Chaidari, Athens, Attica
  - Local Institution - 4810, Kalyftaki-N. Kifissia, Attica
  - Local Institution - 4806, Marousi, Attica
  - Local Institution - 4801, Heraklion
  - Local Institution - 4811, Thessaloniki
- Hungary (8):
  - Local Institution - 4601, Pécs, Baranya
  - Local Institution - 1-13JED893, Szeged, Csongrád megye
  - Local Institution - 4610, Szeged, Csongrád megye
  - Local Institution - 4602, Budapest
  - Local Institution - 4612, Budapest
  - Local Institution - 1-13JED8D1, Gyöngyös
  - Local Institution - 4611, Gyöngyös
  - Local Institution - 4603, Miskolc
- India (6):
  - Local Institution - 7401, Nagpur, Maharashtra
  - Local Institution - 7405, Chandigarh, Punjab
  - Local Institution - 7406, Ajmer, Rajasthan
  - Local Institution - 7403, Hyderabad
  - Local Institution - 7404, Kolkata
  - Local Institution - 7402, Varanasi
- Israel (4):
  - Local Institution - 3101, Jerusalem, Jerusalem
  - Local Institution - 3103, Ashkelon, Tel Aviv
  - Local Institution - 3102, Petah Tikva
  - Local Institution - 3104, Ramat Gan
- Italy (18):
  - Local Institution - 1-140JNJT7, Salerno, Campania
  - Local Institution - 1-13JED80W, Rome, Lazio
  - Local Institution - 2322, Rome, Lazio
  - Local Institution - 1-13JED82O, Rome, Lazio
  - Local Institution - 2320, Rome, Lazio
  - Local Institution - 2301, Rome, Lazio
  - Local Institution - 1-13JED83E, Brescia, Lombardy
  - Local Institution - 2324, Brescia, Lombardy
  - Local Institution - 2304, Milan, Lombardy
  - Local Institution - 2323, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico di Modena, Baggiovara, Modena
  - Local Institution - 2307, Ponderano (Biella), Piedmont
  - Local Institution - 2321, Rome, Roma
  - Local Institution - 2308, Florence, Tuscany
  - Local Institution - 2305, Monza
  - Local Institution - 2302, Pisa
  - Local Institution - 2303, Roma
  - Local Institution - 2309, Roma
- Japan (27):
  - Local Institution - 1-13H98LYW, Iizuka, Fukuoka
  - Local Institution - 7503, Iizuka, Fukuoka
  - Local Institution - 7525, Kōriyama, Fukushima
  - Local Institution - 7522, Sapporo, Hokkaido
  - Local Institution - 7526, Himeji-Shi, Hyōgo
  - Local Institution - 1-13H98LIT, Toride-shi, Ibaraki
  - Memory Clinic Toride, Toride-shi, Ibaraki
  - Local Institution - 7514, Takamatsu, Kagawa-ken
  - Local Institution - 7505, Hadano, Kanagawa
  - Local Institution - 7507, Kawasaki-Shi, Kanagawa
  - Local Institution - 7520, Yokohama, Kanagawa
  - Local Institution - 7502, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Local Institution - 7511, Kyoto, Kyoto
  - Local Institution - 7506, Tsu, Mie-ken
  - Asakayama General Hospital, Sakai, Osaka
  - Local Institution - 7501, Takatsuki, Osaka
  - Local Institution - 7512, Yoshinogawa, Tokushima
  - Local Institution - 7518, Hachiōji, Tokyo
  - Local Institution - 7521, Setagaya-Ku, Tokyo
  - Local Institution - 7519, Setagaya-Ku, Tokyo
  - Local Institution - 7528, Setagaya-Ku, Tokyo
  - Local Institution - 7527, tabashi City, Tokyo
  - Local Institution - 7516, Hiroshima
  - Local Institution - 1-13H98LTZ, Kumamoto
  - Local Institution - 7524, Kumamoto
  - Local Institution - 7523, Tatebayashi
- Mexico (7):
  - Hospital Universitario de Saltillo Dr Gonzalo Valdes Valdes, Saltillo Centro, Coahuila
  - Local Institution - 1504, Zona Urbana Río Tijuana, Estado de Baja California
  - Local Institution - 1507, Zapopan, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey, Nuevo León
  - Local Institution - 1505, Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Local Institution - 1506, México
- Peru (2):
  - Local Institution - 6102, Miraflores, Lima region
  - Local Institution - 6101, Callao
- Poland (15):
  - Centrum Medyczne HCP Szpital im. Jana Pawla II, Poznan, Greater Poland Voivodeship
  - Osrodek Badan Klinicznych Appletreeclinics, Lódz, Lódzkie
  - Uniwersyteckie Centrum Kliniczne w Gdansku - Smoluchowskiego 17, Gdansk, Pomeranian Voivodeship
  - Local Institution - 1-13JAX170, Gdansk, Pomeranian Voivodeship
  - Local Institution - 4215, Iława, Warmian-Masurian Voivodeship
  - Local Institution - 4204, Bydgoszcz
  - Local Institution - 4208, Katowice
  - Local Institution - 4205, Katowice
  - Local Institution - 4213, Kielce
  - Medycyna Milorzab sp. z o.o., Lodz
  - Local Institution - 4214, Lodz
  - NZOZ NEUROMED M. I M. Nastaj Spolka Partnerska -Lublin, Lublin
  - Local Institution - 4209, Siemianowice Śląskie
  - Osrodek Badawczo Naukowo Dydaktyczny Chorób Otepiennych im Ksiedza Henryka Kardynala Gulbinowicza, Ścinawa
  - Local Institution - 4211, Wroclaw
- Portugal (6):
  - Local Institution - 2701, Guimarães, Braga District
  - Local Institution - 2704, Lisbon, Lisbon District
  - Local Institution - 2702, Torres Vedras, Lisbon District
  - Local Institution - 2703, Matosinhos Municipality, Porto District
  - Local Institution - 2705, Lisbon
  - Local Institution - 2706, Lisbon
- Puerto Rico (5):
  - Local Institution - 1303, Bayamón
  - Local Institution - 1301, Bayamón
  - Local Institution - 1305, Carolina
  - Local Institution - 1302, San Juan
  - Barbara Diaz Hernandez MD Research Inc, San Juan
- Romania (5):
  - CMI Dr. Buhas Ramocea Elena Daniela - Cabinet Medical de Psihiarie, Oradea, Bihor County
  - Prof Dr Alexandru Obregia Clinical Psychiatric Hospital- Centrul de Sanatate Mintala, Bucharest
  - Local Institution - 4902, Constanța
  - Local Institution - 4903, Craiova
  - S.C. Carpe Diem SRL, Sibiu
- Serbia (13):
  - Local Institution - 4307, Belgrade, Belgrade
  - Local Institution - 4302, Belgrade, Belgrade
  - Clinical Hospital Center Dragisa Misovic Dedinje, Belgrade
  - Local Institution - 4304, Belgrade
  - Local Institution - 4308, Belgrade
  - Local Institution - 1-13JAX17Q, Gornja Toponica
  - Special Hospital for Psychiatric Diseases "Gornja Toponica", Gornja Toponica
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - Local Institution - 4301, Kragujevac
  - Local Institution - 4310, Kragujevac
  - University Clinical Center Kragujevac, Kragujevac
  - Local Institution - 4309, Novi Sad
  - Local Institution - 4311, Vršac
- Slovakia (7):
  - Univerzitna nemocnica L Pasteura Kosice-Rastislavova 43, Košice, Košice Region
  - MUDr. Beata Dupejova, Neurologicka ambulancia, s.r.o., Banská Bystrica
  - KONZILIUM s.r.o, Dubnica nad Váhom
  - EPAMED s.r.o, Košice
  - Local Institution - 1-13JED85D, Pezinok
  - Psychiatrická nemocnica Philippa Pinela Pezinok, Pezinok
  - Crystal Comfort, s.r.o., Vranov nad Topľou
- South Korea (16):
  - Local Institution - 7208, Buk-gu, Daegu Gwang'yeogsi
  - Local Institution - 7214, Ansan-si, Gyeonggido
  - Local Institution - 7207, Seongnam-si, Gyeonggido
  - Local Institution - 7216, Yongin-si, Gyeonggido
  - Local Institution - 7205, Incheon, Incheon Gwang'yeogsi
  - Local Institution - 7217, Seoul, Seoul Teugbyeolsi
  - Local Institution - 7213, Seoul, Seoul Teugbyeolsi
  - Local Institution - 7210, Seoul, Seoul Teugbyeolsi
  - Local Institution - 7215, Seoul, Seoul Teugbyeolsi
  - Local Institution - 7212, Yeongdeungpo-gu, Seoul Teugbyeolsi
  - Local Institution - 7218, Gangwon-do
  - Local Institution - 7202, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Local Institution - 7203, Seoul
  - Local Institution - 7201, Seoul
  - Hanyang University Seoul Hospital, Seoul
- Spain (11):
  - Local Institution - 2211, Majadahonda, Madrid
  - Local Institution - 2213, Málaga, Málaga
  - Local Institution - 2205, Barcelona
  - Local Institution - 2212, Lleida
  - Local Institution - 2207, Madrid
  - Local Institution - 2210, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Local Institution - 2201, Seville
  - Hospital Universitario Rio Hortega, Valladolid
  - Local Institution - 2202, Zamora
  - Hospital Viamed Montecanal, Zaragoza
- Turkey (Türkiye) (6):
  - Local Institution - 4702, Atakum, Samsun
  - Local Institution - 4706, Ankara
  - Local Institution - 4701, Eskişehir
  - Local Institution - 4704, Istanbul
  - Local Institution - 4705, Izmir
  - Local Institution - 4703, Izmir
- United Kingdom (9):
  - Local Institution - 2110, Ilford, Greater London
  - Local Institution - 2108, Swinton, Greater Manchester
  - Local Institution - 2105, Aberdeen
  - Local Institution - 2109, Chertsey
  - Local Institution - 2106, Leeds
  - Local Institution - 2104, Motherwell
  - Local Institution - 2111, Preston
  - Local Institution - 2107, Sheffield, SouthYorkshire
  - Local Institution - 2103, Swindon

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05980949.html